CLINICAL TRIAL: NCT02248194
Title: Tactile Versus Hysteroscopic Electrosurgical Ablation in Cases of Dysfunctional Uterine Bleeding
Brief Title: Tactile Electrosurgical Ablation in Cases of Dysfunctional Uterine Bleeding
Acronym: TEA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mostafa Hussein (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Mostafa Hussein, Dr, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tactile ablation
Record Dates: First submitted 2014-01-22; First posted 2014-09-25 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Dysfunction Uterine Bleeding
Keywords: Dysfunction uterine bleeding; Hysteroscopic endometrial ablation; Tactile endometrial ablation; Hysteroscopic difficulties; Quality of life; Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1"Tactile electrosurgical ablation" (Experimental): Endometrial ablation will be done by Tactile electrosurgical ablation probe.
  Interventions: Device: Hysteroscopic endometrial ablation
- Group 2 "Hysteroscopic endometrial ablation" (Active Comparator): Hysteroscopic endometrial ablation will be done by trans-cervical resection of endometrium.
  Interventions: Device: Tactile electrosurgical ablation probe

INTERVENTIONS:
Device: Tactile electrosurgical ablation probe
  Arms: Group 2 "Hysteroscopic endometrial ablation"
Device: Hysteroscopic endometrial ablation
  Other Names: Transcervical resection of the endometrium
  Arms: Group 1"Tactile electrosurgical ablation"

SUMMARY:
Abnormal uterine bleeding (AUB) is any alteration in the pattern or volume of menstrual blood ﬂow and heavy menstrual bleeding affects up to 30% of women at some time during their reproductive years. Abnormal menstruation can be due to conditions such as pregnancy complication uterine fibroids and adenomyosis, but in a large proportion of cases, the etiology is unclear, a condition generally referred to as dysfunctional uterine bleeding (DUB). Treatment options for DUB include symptomatic medical treatment or surgery, traditionally hysterectomy.

Hysteroscopically guided endometrial ablation methods have been shown to be effective and safe alternatives to hysterectomy for management of DUB. These methods require particular skills and experience and a long learning curve to be performed effectively and safely.

Through the past three decades DUB patients in Assiut university hospital were treated with either electrosurgical ablation or hysterectomy. When faced with hysteroscopic challenges during transcervical resection of the endometrium or rollerball coagulation, we used to shift to thermal balloon as backup method . However, expensive uterine balloon could not infrequently be afforded because of financial constrains and limited health resources . Therefore, another method was used as backup for hysteroscopic failures. It was first tried via insulating the conventional double-ended uterine curette then through a specially designed tactile electrosurgical ablation (TEA) probe.The technique of TEA is largely similar to the dilatation and curettage procedure both principally and practically. Hence, the basic requirements for its performance are the general awareness with electrosurgical principles and adequate experience in performing dilatation and curettage. TEA is done by specially designed tactile diathermy probe that carried the job of electrosurgical ablation without hysteroscopy or distension media first in an experimental session that clearly clarified the reproducibility of the depth of thermal damage and safety of the tactile electrosurgical ablator . Thereafter, TEA was successfully performed with satisfactory short and medium term outcomes for ten cases with DUB during an active, relentless bleeding attack. TEA is done under laparoscopic monitoring.

The aim of the present work is to present TEA as a simple, inexpensive, novel backup approach for treatment of DUB.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dysfunctional uterine bleeding aged between 40 to 50 years
* Unsuccessful medical treatment.
* No intrauterine abnormalities.
* Endometrial biopsy negative for atypia and cancer.
* follicle stimulating hormone level not exceeds 30 mills-International unit
* Family complete
* Patients who are not candidate for hysterectomy because of medical or surgical risks.

Exclusion Criteria:

* Coexisting gynecological pathology (e.g. uterovaginal prolapsed, ovarian pathology, pelvic inflammatory disease, cervical atypia).
* Endometrial hyperplasia with atypia and cancer..
* History or evidence of malignancy.
* Hyperplasia in the endometrial biopsy.
* Uterine size more than 12 weeks in size.
* Women with caesarean or myomectomy scar

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2010-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the treatment at 12 month follow up | 12 moth
  Satisfaction with the treatment will be measured at 1 year post procedure on 3-point scale-very satisfied, satisfied, and not satisfied.
Change in menstrual status. | At 3, 6, 9, and12 months pot operatve.
  Menstrual status will be reported as
  * Normal menstrual flow.
  * Light menstrual bleeding.
  * Heavy menstrual bleeding.
  * The need for hysterectomy.

SECONDARY OUTCOMES:
Acceptability of treatment | 4 weeks
  Acceptability of the procedure will be assessed in 3- point scale as cure or acceptable improvement in symptoms, treatment acceptable and would recommend treatment to others or not acceptable
Changes in health related quality of life | At 3, 6, 9, and 12 months post operative.
  Health-related quality of life parameters will be completed using
  * Short form-12 (SF12).
  * Life style questionnaires including Work affection will be measured by the number of days absence from the work due to menses as following, non ,non but work suffer, 1 day and >2 days.
  * sexual life affection will be measured in two point as no or yes.
Difference in operative time between the two groups in minutes. | 0-60 minutes
  Difference in operative time is calculated using a stop watch.The zero minute is the time of starting the procedure. The stop watch is on at the zero minute then sopped at the end of the procedure.time of anesthesia is not included.
Reporting of any intro-operative complications. | 0-60 minutes.
  Intro-operative complications includes
  * Cervical laceration.
  * Perforation of the uterus.
  * Hemorrhage
  * Fluid overload.
Reporting of any technical complications. | 0-60 minutes
  Technical complications for transcervical resection of the endometrium (TCRE) includes
  * Poor uterine distention.
  * Slow clearance of the debris.
  * Inefficient cutting.
  * Poor visualization.
  * problem of diathermy.
  * Problems with the camera.
  * problems with light source.
  Technical complications for tactile electrosurgical ablation (TEA) includes
  * Insulation problem.
  * Connection problem.
  * Inefficient diathermy power.
Difference in post-operative pain score using visual analogue scale between the two groups. | 4 hours.
  Difference in post-operative pain score using visual analogue scale from 1-10.
Time needed for post operative recovery (days) of pain, vaginal bleeding, vaginal discharge, till full recovery and till return to work. | 28 days post operative
Length of hospital stay in days | up to 2 days
  Length of hospital stay in days is calculated from the day of operation till day of discharge.
Difference in the cost of the two surgical procedure. | up to one hour.
  Direct cost of the surgical procedure itself is calculated.The cost of the TCRE procedure will include the cost paid for the hysteroscopic unit and the cost of glycine used as distension media.The cost of the TEA procedure will include the cost of laparoscopy, the cost of TEA probe, and the cost of diagnostic hysteroscopy. The cost of the investigations, anesthesia, pre and post operative treatments will be excluded from analysis as they are the same for both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Woman's Health Hospital-Assiut University., Asyut, Egypt